CLINICAL TRIAL: NCT04212598
Title: The Value of Sintilimab Consolidation Therapy After Definitive Concurrent Chemoradiotherapy for Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma, an Open, Prospective, Single-arm Phase II Study
Brief Title: The Value of Sintilimab Consolidation Therapy After Definitive Concurrent Chemoradiotherapy for Locally Advanced Thoracic Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Conghua Xie,MD,PhD, Director, Head of Radiation and Medical Oncology, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immune consolidation therapy
Record Dates: First submitted 2019-12-21; First posted 2019-12-27 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Chemoradiotherapy; Esophageal Squamous Cell Carcinoma; Immunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: This is a single arm phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Definitive concurrent chemoradiotherapy or radiotherapy arm (Experimental): Patients who completed concurrent chemoradiotherapy standard dose would received the Sintilimab as a consolidate therapy for one year.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Patients who completed concurrent chemoradiotherapy standard dose would received the Sintilimab as a consolidate therapy for one year.

SUMMARY:
Esophageal cancer is a kind of disease with high incidence and mortality. Definitive concurrent chemoradiotherapy is an important treatment for locally advanced esophageal squamous cell carcinoma. To Investigate the value of immunotherapy consolidation in locally advanced esophageal squamous cell carcinoma after completing radical concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
In East countries, especially China, more than 75 percent of esophageal cancers are primary squamous cell cancers located in the middle and upper thoracic segments, whereas adenocarcinoma accounted for less than 20 percent.Unlike other malignancies, more than half of esophageal cancer were diagnosed as locally advanced at the time of diagnosis. Definitive concurrent chemoradiotherapy is an important treatment for locally advanced esophageal squamous cell carcinoma.

Immune checkpoint inhibitors are a new class of antitumor drugs. They are different from traditional cytotoxic chemotherapy drugs and can target the regulatory molecules that play an inhibitory role in the tumor immune system.

Recent clinical studies had shown that for locally advanced non-small cell lung cancer, maintenance therapy with the immune checkpoint inhibitor could significantly improve the overall survival for locally advanced non-small cell lung cancer after definitive concurrent chemoradiotherapy. Moreover, the immune checkpoint inhibitor PD-1 has also been shown to be a promising anticancer agent in esophageal cancers. Therefore, the present study intended to give a standard dose (50.4Gy/28F) to locally advanced esophageal squamous cell carcinoma for radical chemoradiotherapy, and than to give the Sintilimab as consolidation therapy for 1 year after completion of radiotherapy. At the time point of 6 weeks after radiotherapy, all participates need a full evaluation of the treatment response. In patients with residual disease, we would give them an additional radiotherapy boost to 61.2 Gy/34F under the guidance of PET-CT or ultrasound endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1; Life expectancy >6 months;
* Stage II/III esophageal cancer;
* Pathology confirmed squamous cell carcinoma;
* Hemoglobin ≥10g/dl, WBC ≥3.0 x 109/L, platelet ≥100 x 109/L; CR≤ 1.0x normal upper limit, total bilirubin ≤ 1.5x normal upper limit, AST and ALT≤ 1.5x normal upper limit, AKP≤ 2.5x normal upper limit;
* Have a full understanding of this study, participate voluntarily, have follow-up conditions and sign the informed consent;

Exclusion Criteria:

* Stage IV esophageal cancer;
* Esophageal adenocarcinoma;
* Gastric esophageal junction adenocarcinoma;
* ECOG > 2;
* Progression after first-course radiotherapy;
* Existing active infection, such as active tuberculosis, hepatitis, etc.;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-11-03 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with disease progression within 2 years after treatment | 2-years
  Progression-free survival is measured from the date of enrolling to the date of disease progression or death from any cause or final follow-up

SECONDARY OUTCOMES:
Percentage of patients who died within 2 years after treatment | 2-years
  Progression-free survival is measured from the date of enrolling to the date of death from any cause or final follow-up

OTHER OUTCOMES:
The number of patients with treatment-related toxicity between the treatment period and half a year after treatment | 0.5-year
  Acute toxicities were scored according to the Common Toxicity Criteria for Adverse Events, version 3.0 (National Cancer Institute, NCI, Rockville, MD).

CONTACTS AND LOCATIONS:
Overall Officials: Conghua Xie, MD, Study Director — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Background] Suh YG, Lee IJ, Koom WS, Cha J, Lee JY, Kim SK, Lee CG. High-dose versus standard-dose radiotherapy with concurrent chemotherapy in stages II-III esophageal cancer. Jpn J Clin Oncol. 2014 Jun;44(6):534-40. doi: 10.1093/jjco/hyu047. Epub 2014 Apr 24. PMID 24771865
- [Background] Zhang Z, Liao Z, Jin J, Ajani J, Chang JY, Jeter M, Guerrero T, Stevens CW, Swisher S, Ho L, Yao J, Allen P, Cox JD, Komaki R. Dose-response relationship in locoregional control for patients with stage II-III esophageal cancer treated with concurrent chemotherapy and radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Mar 1;61(3):656-64. doi: 10.1016/j.ijrobp.2004.06.022. PMID 15708243